CLINICAL TRIAL: NCT00171613
Title: A Study of Octreotide Depot vs Saline Control in Pediatric Hypothalamic Obesity Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSMS995B2403E1
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Hypothalamic Obesity
Keywords: Obesity
MeSH Terms: conditions — Sexual Infantilism; Obesity | interventions — Octreotide

INTERVENTIONS:
Drug: Octreotide

SUMMARY:
The extension protocol is designed to allow those patients randomized to placebo in the core portion of the protocol to receive a 6 month treatment of open label octreotide and allow those patients randomized to octreotide who appeared to benefit from treatment, to continue to receive octreotide.

ELIGIBILITY:
Inclusion Criteria

- Patient must provide written informed consent

Exclusion Criteria

* Any patient that experienced unresolved safety complications at any time during the original protocol CSMS995B2403
* Patients with a history of gallstones or any patient developing gallstones during the course of the core protocol
* Patients for whom there are safety or tolerability concerns for continuing Octreotide Depot
* Any patient requiring additional treatment for their original cranial insult related to cranial trauma, or to tumor recurrence or its treatment Refer to the original protocol for details of inclusion & exclusion criteria. Any patient granted a waiver to participate in the core protocol will be allowed to continue to participate in the extension protocol.

Other protocol-defined inclusion / exclusion criteria may apply.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32
Dates: Start 2005-02; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in BMI

SECONDARY OUTCOMES:
Change from baseline in weight, leptin, insulin AUC, C-peptide AUC, amylin AUC, glucose AUC, dietary intake, physical activity, waist-to-hip ratio, visceral and subcutaneous abdominal fat

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis